CLINICAL TRIAL: NCT00079729
Title: Directly Observed Therapy (DOT) in HIV-Infected Adolescents: Part A-Focus Groups
Brief Title: Directly Observed Therapy in HIV Infected Adolescent Focus Groups
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: PACTG P1036A; 10193 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2004-03-11; First posted 2004-03-12 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to help researchers use information from HIV infected adolescents to design a directly observed therapy (DOT) program that will help adolescents take their anti-HIV medications correctly.

DETAILED DESCRIPTION:
The rate of HIV infection among adolescents is increasing at an alarming rate. Adherence to antiretroviral therapy has been a major challenge in achieving and maintaining adequate control of the disease in this population. DOT has been shown effective in individuals with tuberculosis (TB), but DOT in HIV infected populations has not been thoroughly examined. This study will collect information from HIV infected adolescents in order to establish a DOT program that will increase successful adherence to HIV treatment and will benefit the public by preventing development of viral resistance and reducing the risk of transmission.

Adolescent participants in this study will be assigned to one of three 2-hour focus group sessions, each at a different site. The participants will complete a questionnaire and will give input about designing a DOT intervention model that will be accepted by adolescents. The model will then be used in a pilot study to determine the feasibility of implementing DOT programs in the community to help HIV infected adolescents.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected due to high-risk behavior
* Regular attendee of local adolescent HIV support group
* Current use of antiretrovirals or history of antiretroviral therapy
* Permission of parent or legal guardian if participant is less than the legal age of consent. Assent of the minor participant should be obtained where required.

Exclusion Criteria:

* Perinatal HIV infection
* Visibly distraught or emotionally unstable
* Pregnancy or breast-feeding

Ages: 16 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30
Dates: Start 2004-04; Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Flynn, MD, Study Chair — St. Jude Children's Research Hospital
Locations (3):
- United States (3):
  - Los Angeles County Medical Center/USC, Los Angeles, California
  - University of Miami (Pediatric), Miami, Florida
  - St. Jude Childrens Research Hospital, Memphis, Memphis, Tennessee

REFERENCES:
- [Background] Murphy DA, Wilson CM, Durako SJ, Muenz LR, Belzer M; Adolescent Medicine HIV/AIDS Research Network. Antiretroviral medication adherence among the REACH HIV-infected adolescent cohort in the USA. AIDS Care. 2001 Feb;13(1):27-40. doi: 10.1080/09540120020018161. PMID 11177463
- [Background] Babudieri S, Aceti A, D'Offizi GP, Carbonara S, Starnini G. Directly observed therapy to treat HIV infection in prisoners. JAMA. 2000 Jul 12;284(2):179-80. doi: 10.1001/jama.284.2.179. No abstract available. PMID 10889588
- [Background] Lanzafame M, Trevenzoli M, Cattelan AM, Rovere P, Parrinello A. Directly observed therapy in HIV therapy: A realistic perspective? J Acquir Immune Defic Syndr. 2000 Oct 1;25(2):200-1. doi: 10.1097/00042560-200010010-00018. No abstract available. PMID 11103053
- [Background] Mitty JA, McKenzie M, Stenzel M, Flanigan T, Carpenter CC. Modified directly observed therapy for treatment of human immunodeficiency virus. JAMA. 1999 Oct 13;282(14):1334. doi: 10.1001/jama.282.14.1334. No abstract available. PMID 10527179
- [Result] Garvie PA, Lawford J, Flynn PM, Gaur AH, Belzer M, McSherry GD, Hu C; Pediatric AIDS Clinical Trials Group 1036A Study Team. Development of a directly observed therapy adherence intervention for adolescents with human immunodeficiency virus-1: application of focus group methodology to inform design, feasibility, and acceptability. J Adolesc Health. 2009 Feb;44(2):124-132. doi: 10.1016/j.jadohealth.2008.05.006. Epub 2008 Oct 18. PMID 19167660